CLINICAL TRIAL: NCT06609005
Title: A Phase 1 and Phase 2, Multi-Center, Open-Label Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Evidence of Antitumor Activity of INV-9956 in Adult Patients With Advanced Metastatic Castration Resistant Prostate Cancer
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of INV-9956 in Adult Patients With Advanced Metastatic Castration Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Ionova Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INV-9956-101
Record Dates: First submitted 2024-09-11; First posted 2024-09-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Advanced Metastatic Castration Resistant Prostate Cancer
Keywords: mCRPC; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase 1 INV-9956 Dose escalation Dose level 1 (Experimental): INV-9956 Dose escalation Dose level 1 is co-administered with dexamethasone and fludrocortisone acetate
  Interventions: Drug: INV-9956
- Phase 1 INV-9956 Dose escalation Dose level 2 (Experimental): INV-9956 Dose escalation Dose level 2 is co-administered with dexamethasone and fludrocortisone acetate
  Interventions: Drug: INV-9956
- Phase 1 INV-9956 Dose escalation Dose level 3 (Experimental): INV-9956 Dose escalation Dose level 3 is co-administered with dexamethasone and fludrocortisone acetate
  Interventions: Drug: INV-9956
- Phase 2 INV-9956 Dose expansion - Cohort A (Experimental): INV-9956 is co-administered with dexamethasone and fludrocortisone acetate
  Interventions: Drug: INV-9956
- Phase 2 INV-9956 Dose expansion - Cohort B (Experimental): INV-9956 is co-administered with dexamethasone and fludrocortisone acetate
  Interventions: Drug: INV-9956
- Phase 1 INV-9956 Dose escalation beyond the optimal dose - Dose level 4 (Experimental): INV-9956 Dose escalation Dose level 4 is co-administered with dexamethasone and fludrocortisone acetate
  Interventions: Drug: INV-9956
- Phase 1 INV-9956 Dose escalation beyond the optimal dose - Dose level 5 (Experimental): INV-9956 Dose escalation Dose level 5 is co-administered with dexamethasone and fludrocortisone acetate
  Interventions: Drug: INV-9956
- Phase 1 INV-9956 Dose escalation beyond the optimal dose - Dose level 6 (Experimental): INV-9956 Dose escalation Dose level 6 is co-administered with dexamethasone and fludrocortisone acetate
  Interventions: Drug: INV-9956

INTERVENTIONS:
Drug: INV-9956 — INV-9956 is co-administered with dexamethasone and fludrocortisone acetate

SUMMARY:
This is a Phase 1 and Phase 2 study to evaluate the safety and antitumor activity of INV-9956 in adult patients with advanced metastatic Castration Resistant Prostate Cancer.

DETAILED DESCRIPTION:
This is a Phase 1 and Phase 2 study to evaluate the safety and antitumor activity of INV-9956 in adult patients with advanced metastatic Castration Resistant Prostate Cancer.

The entire study consists of two parts: Phase 1 for dose escalation and Phase 2 for dose expansion.

Phase 1 dose escalation of INV-9956 follows a real time monitored, PK/PD and safety guided scheme with a traditional 3+3 design for DLT assessment.

Phase 2 aims to reassure the safety profile and better define efficacy. Phase 2 consists of up to 2 cohorts by different AR gene status:

* Cohort A: AR mutant CRPC
* Cohort B: AR wide-type CRPC (optional) Currently enrolling patients under Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained.
2. Male aged ≥ 18 years.
3. Histologically confirmed adenocarcinoma of the prostate.
4. Castration resistant prostate cancer with serum testosterone <50 ng/dL.
5. Metastatic disease.
6. Ongoing androgen deprivation therapy with GnRH analogue or antagonist, or have had bilateral orchiectomy.
7. Received at least one prior line of taxane-based chemotherapy and at least one line of hormonal AR targeted therapy (eg, abiraterone, enzalutamide). Patients who have refused or were intolerant to taxane-based chemotherapy may be enrolled.
8. ECOG performance status 0-1.
9. Adequate marrow, liver and kidney function.
10. INR ≤1.5.
11. Able to swallow study treatment.
12. Has a life expectancy of > 3 months.

Exclusion Criteria:

1. Have a medical condition such as Crohn's disease or have undergone significant surgery to the gastrointestinal tract that could impair absorption or that could result in short bowel syndrome with diarrhea due to malabsorption.
2. History of pituitary or adrenal dysfunction.
3. Poorly controlled diabetes mellitus.
4. Clinically significant abnormality in serum potassium and sodium.
5. Have a serious nonmalignant disease (eg, hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
6. Active or unstable cardio-/cerebro-vascular disease, including thromboembolic events.
7. History of congestive heart failure; cardiac disease, myocardial infarction within 6 months prior to enrollment.
8. Prolonged QTcF interval.
9. Active infection or other medical condition that would make corticosteroid contraindicated.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2028-01-17 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum tolerated dose (MTD) | Within first 28 days of treatment
  The highest dose level at which at least 6 patients have been treated and less than 33% of patients experienced a DLT.
Phase 1: Recommended dose range (RDR) | 12 months
  The RDR will be determined based on the PK and PD data, the preliminary clinical activity of INV-9956, as well as the incidence rate and nature of the toxicities observed in subsequent cycles beyond Cycle 1
Phase 2: Evaluate Radiographic progression-free survival (rPFS) | 12 months
  To evaluate rPFS per PCWG-modified RECIST v1.1 (soft tissue response) and PCWG3 criteria (bone metastases)
Phase 2: Evaluate overall response rate (ORR) | 12 months
  To evaluate ORR per PCWG-modified RECIST v1.1 (soft tissue response) and PCWG3 criteria (bone metastases)

SECONDARY OUTCOMES:
Phase 1: Characterize the safety of INV-9956 as assessed by CTCAE v5.0 | 12 months
  To analyze the safety profile of INV-9956 as a single agent by AE, clinical lab test results, ECG and Vital signs changes
Phase 1: Determine the PK using AUC of INV-9956 | 12 months
  To determine the pharmacokinetics (PK) using AUC of INV-9956 after a single dose and at steady state after multiple doses
Phase 1: Determine the PK using Cmax of INV-9956 | 12 months
  To determine the pharmacokinetics (PK) using Cmax of INV-9956 after a single dose and at steady state after multiple doses
Phase 1: Determine the blood concentration of steroid hormone | 12 months
  To determine the blood concentration of steroid hormones at various timepoints as PD markers for INV-9956
Phase 1: Evaluate Radiographic progression-free survival (rPFS) | 12 months
  To evaluate rPFS per PCWG-modified RECIST v1.1 (soft tissue response) and PCWG3 criteria (bone metastases)
Phase 1: Evaluate overall response rate (ORR) | 12 months
  To evaluate ORR per PCWG-modified RECIST v1.1 (soft tissue response) and PCWG3 criteria (bone metastases)
Phase 2: Characterize the safety of INV-9956 as assessed by CTCAE v5.0 | 12 months
  To analyze the safety profile of INV-9956 as a single agent by AE, clinical lab test results, ECG and Vital signs changes
Phase 2: Determine the PK using AUC of INV-9956 | 12 months
  To determine the pharmacokinetics (PK) using AUC of INV-9956 after a single dose and at steady state after multiple doses
Phase 2: Determine the PK using Cmax of INV-9956 | 12 months
  To determine the pharmacokinetics (PK) using Cmax of INV-9956 after a single dose and at steady state after multiple doses
Phase 2: Determine the blood concentration of steroid hormone | 12 months
  To determine the blood concentration of steroid hormones at various timepoints as PD markers for INV-9956

CONTACTS AND LOCATIONS:
Locations (17):
- United States (7):
  - Honor Health, Scottsdale, Arizona
  - Hoag Family Cancer Institute, Newport Beach, California
  - UC Irvine Medical Center, Orange, California
  - Next Oncology - Houston, Houston, Texas
  - UT Health, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia
  - Summit Cancer Centers, Spokane, Washington
- China (10):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - He'nan Cancer Hospital, Zhengzhou, He'Nan
  - Hu'nan Cancer Hospital, Changsha, Hu'Nan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shandong Cancer Hospital, Ji'nan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No